CLINICAL TRIAL: NCT00078091
Title: Bardet-Biedl Syndrome: Phenotype and Metabolic Characteristics
Brief Title: Genetics and Clinical Characteristics of Bardet-Biedl Syndrome
Status: Terminated | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040123; 04-HG-0123
Record Dates: First submitted 2004-02-18; First posted 2004-02-19 (Estimated); Last update posted 2019-12-04 (Actual); Status verified 2016-02-05

CONDITIONS: Bardet-Biedl Syndrome
Keywords: Obesity; Retinopathy; Dyslipidemia; Insulin Resistance; Hypogonadism; Polydactyly; Bardet-Biedl Syndrome; BBS
MeSH Terms: conditions — Bardet-Biedl Syndrome; Obesity; Retinal Diseases; Dyslipidemias; Insulin Resistance; Hypogonadism; Polydactyly

SUMMARY:
This study will evaluate patients with a rare inherited condition called Bardet-Biedl syndrome . The purpose of the study is to learn more about the genetics and clinical characteristics of this disorder. Patients may have the following problems: polydactyly (extra fingers and toes); retinal dystrophy (changes in the retina that may lead to vision problems, including blindness); obesity and diabetes (overweight and high blood sugar due to failure of body organs to respond to insulin); cognitive dysfunction (difficulties with learning and understanding); hypogenitalism (decreased functioning of the ovaries in women and the testes in men); kidney anomalies (changes in the structure or function of the kidneys); heart disease; and hepatic fibrosis (liver disease).

Patients with Bardet-Biedl syndrome may be eligible for this study. First-degree relatives will also be enrolled for certain tests and procedures. Candidates are screened with a review of their medical records, laboratory tests, and x-rays.

Patients in this study undergo the following tests and procedures:

* Medical and family history and physical examination, including body measurements.
* Blood tests to evaluation kidney, liver, heart, and hormonal function, and for genetic studies and other research purposes.
* Dual emission x-ray absorptiometry (DEXA) scan to measure the amount of total body fat. For this test, the subject lies on a table for scanning with low-dose X-rays.
* Computed tomography (in adults) of the abdomen to measure abdominal fat. CT uses a small amount of radiation to obtain images of internal body structures.
* Magnetic resonance imaging (in children) of the abdomen to measure abdominal fat. MRI uses a magnetic field and radio waves to obtain images of internal body structures.
* Oral glucose tolerance tests to measure blood glucose and insulin levels. For this test, the patient drinks a glucose (sugar) solution. Blood samples are drawn through an IV catheter before the test begins and at 1, 2, and 3 hours after drinking the solution.
* Complete eye examination to look for retinal changes and to assess vision, and, if medically needed, an examination of the ear, nose, and throat to check for hearing and breathing abnormalities.
* Tests of learning ability in patients over 5 years of age. For younger patients, a parent is asked about the child's development.
* Ultrasound study of the ovaries and uterus in females and of the testes in males.
* Photographs of the face, hands, feet, body, and genitalia, if the patient agrees.
* Meeting with investigators and a genetic counselor for review of test findings when the studies are completed.

Relatives of patients have a complete medical and family history and physical examination. Blood is drawn for assessment of kidney, liver, heart, and hormonal function and for genetic study and other research purposes. Relatives over 5 years of age may have tests of learning ability and cognition. For younger patients, a parent is asked about the child's development. Relatives meet with investigators and a genetic counselor for review of test findings when the studies are completed.

DETAILED DESCRIPTION:
Although the Bardet-Biedl syndrome (BBS: severe obesity, polydactyly, learning disabilities, retinopathy, renal disease and cardiac malformations) was described more than 80 years ago, it is only over the past few years that extensive data on the natural history and molecular pathogenesis of this complex disorder have been reported. We now know that BBS can be caused by mutations in at least 12, genes and, although it is typically inherited in an autosomal recessive pattern, BBS may occasionally exhibit more complex inheritance. In this study, we are defining the physical (body mass, percent and distribution of body fat) and metabolic (hyperglycemia, hyperinsulinemia, serum levels of lipids and adipokines) characteristics of glucose and fat metabolism in a cohort of adult and pediatric patients with BBS. We are also characterizing the hypogenitalism in BBS, and attempting to determine its relationship, if any, to the incidence of obesity in BBS. In addition, we are studying the retinal dystrophy, the renal dysfunction, and the nature of the reported mental retardation/learning disability that is found in many patients. We plan to correlate the phenotypic manifestations in our subjects with the results of our mutation analysis studies. Our objective is to learn more about the genetic alterations that may underlie the obesity and associated organ dysfunction that characterizes BBS.

ELIGIBILITY:
* INCLUSION CRITERIA:

We are using the previously published clinical diagnostic criteria for BBS(21) to determine study eligibility of probands. As outlined in that report, we are including patients who present with four of the five primary features or three primary features and two secondary features. Parents are also enrolled for genetic studies. We are not enrolling unaffected siblings or recruiting control subjects, instead, results of testing are being compared to previously published data obtained from appropriate non-BBS control subjects.

The initial determination of eligibility is made by review of prior clinical records. Some patients are not characterized in sufficient detail to know if the person meets the clinical criteria, yet we may suspect the diagnosis. In those cases, the subjects are brought to NIH and undergo clinically appropriate testing to make the diagnosis. If that clinical testing does not confirm the diagnosis, the patient or parents are given appropriate clinical counseling and returned to the care of their personal physician. If features later develop that allow the diagnosis to be made, they may re-enroll and undergo further evaluation.

Our study population includes patients of all ages and ethnic groups, and both genders. The inclusion of children is essential to a research study that is correlating genotype with phenotype, and is attempting an early identification of metabolic abnormalities that may be best treated at an early age. Many of the age-dependent manifestations of BBS develop during childhood and the average age of diagnosis is 9.2 years. Pregnant women and children under the age of 5 yr do not undergo invasive research procedures (i.e. phlebotomy) or procedures involving ionizing radiation (i.e. X-rays or DEXA scans) unless that procedure would be performed as part of standard medical care.

Because cognitive dysfunction is known to be a component of BBS, some patients with impaired cognition and understanding may be evaluated under this protocol. If the investigators believe that an adult patient may not be competent to give informed consent to participate, or does not understand the consent document and the procedures of the study, that patient may be excluded from participation. We may request that the patient and accompanying caregiver also be interviewed by an independent ethics panel to confirm that he or she is competent to give consent and to participate if the team feels this would be useful.

EXCLUSION CRITERIA:

Neither healthy volunteers unrelated to an affected patient nor lab personnel will be enrolled.

We will make efforts to obtain consent from all parents/guardians of minor subjects (i.e. we would not allow a single parent to consent a child when both parents have parental rights). If a single parent or guardian has sole custody/legal responsibility for a child (e.g., a divorce with full custody to one parent or one parent is deceased), we will accept consent from one parent.

Both mothers and fathers of children with BBS (who are also typically enrolled in our protocol, as described above) are eligible to participate in the interview portion of the study. We hypothesize that mothers and fathers will, as groups, have slightly different experiences with coping with courtesy stigma, although a couple may have convergent beliefs, coping mechanisms, and experiences. As such, we predict that we will initially conduct interviews with both parents of the same proband (assuming both parents are interested in participating), although we may target either mothers or fathers only following interim analysis of the interview transcripts.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2004-02-17; Study Completion 2016-02-05

CONTACTS AND LOCATIONS:
Overall Officials: Leslie G Biesecker, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Green JS, Parfrey PS, Harnett JD, Farid NR, Cramer BC, Johnson G, Heath O, McManamon PJ, O'Leary E, Pryse-Phillips W. The cardinal manifestations of Bardet-Biedl syndrome, a form of Laurence-Moon-Biedl syndrome. N Engl J Med. 1989 Oct 12;321(15):1002-9. doi: 10.1056/NEJM198910123211503. PMID 2779627
- [Background] Katsanis N, Ansley SJ, Badano JL, Eichers ER, Lewis RA, Hoskins BE, Scambler PJ, Davidson WS, Beales PL, Lupski JR. Triallelic inheritance in Bardet-Biedl syndrome, a Mendelian recessive disorder. Science. 2001 Sep 21;293(5538):2256-9. doi: 10.1126/science.1063525. PMID 11567139
- [Background] Slavotinek AM, Searby C, Al-Gazali L, Hennekam RC, Schrander-Stumpel C, Orcana-Losa M, Pardo-Reoyo S, Cantani A, Kumar D, Capellini Q, Neri G, Zackai E, Biesecker LG. Mutation analysis of the MKKS gene in McKusick-Kaufman syndrome and selected Bardet-Biedl syndrome patients. Hum Genet. 2002 Jun;110(6):561-7. doi: 10.1007/s00439-002-0733-3. Epub 2002 May 9. PMID 12107442